CLINICAL TRIAL: NCT03447093
Title: The Oral Microbiota in Autoimmune Thyroiditis is Distinctive And Predictive
Brief Title: The Oral Microbiota is Associated With Autoimmune Thyroiditis
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: First Affiliated Hospital of Harbin Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: Yunwei Wei 2017 -12-23
Record Dates: First submitted 2018-02-08; First posted 2018-02-27 (Actual); Last update posted 2018-02-27 (Actual); Status verified 2017-12

CONDITIONS: Microbiota
Keywords: oral microbiota; 16S rRNA gene; Graves' disease; Methimazole; Propylthiouracil; Hashimoto's thyroiditis
MeSH Terms: conditions — Graves Disease; Hashimoto Disease | interventions — Methimazole; Propylthiouracil

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (4):
- Control group: 30 healthy volunteers were included in the healthy control group
- Drug treatment group: 30 GD patients who received treatment with Methimazole Pill or propylthiouracil pill
  Interventions: Drug: Methimazole Pill; Drug: Propylthiouracil Pill
- Incipient group: 30 untreated GD patients
- Hashimoto's thyroiditis group: 30 HT patients

INTERVENTIONS:
Drug: Methimazole Pill — Patients who developed GD received methimazole treatment
  Groups: Drug treatment group
Drug: Propylthiouracil Pill — Patients who developed GD received propylthiouracil treatment
  Groups: Drug treatment group

SUMMARY:
Autoimmune thyroiditis (AITD) mainly includes Hashimoto's thyroiditis (HT) and Grave's disease (GD). Studies have shown that autoimmune thyroiditis is closely related to microbial disorders such as autoimmune thyroiditis However, there is no report on the relationship between oral microecology and autoimmune thyroiditis. Therefore, our group will study the correlation between oral microbiota and AITD.

DETAILED DESCRIPTION:
Autoimmune thyroiditis (AITD) mainly includes Hashimoto's thyroiditis (HT) and Grave's disease (GD). Studies have shown that autoimmune thyroiditis is closely related to microbiological disorders. Intestinal microelements Both ecology and oral microecology belong to the category of microorganisms. It has been reported in the literature that intestinal microecology occurs disorder of autoimmune thyroiditis. However, there is no report on the correlation between oral microecology and autoimmune thyroiditis. When oral microbe flora When the immune system is disrupted, the immune balance is broken, the immune system is over-active, and the autoimmune disease (AID) is lost to the autoantigens and non-pathogenic commensal microbial flora antigens, including rheumatoid arthritis, Sjogren's syndrome, systemic lupus erythematosus, inflammatory bowel disease, and allergic diseases. However, the association between oral microbial flora and AITD remains unclear. . Therefore, the research group will carry out the correlation between oral microbial flora and AITD.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 to 65 years
* GD was clinical diagnosed and thyroid function returned to normal
* HT was clinical diagnosed and thyroid function is normal.

Exclusion Criteria:

* Pregnancy
* Lactation
* Cigarette smoking
* Alcohol addiction
* Hypertension
* Diabetes mellitus
* Lipid dysregulation
* BMI > 27
* Recent (< 3 months prior) use of antibiotics, probiotics, prebiotics, symbiotics, hormonal medication, laxatives, proton pump inhibitors, insulin sensitizers or Chinese herbal medicine
* History of disease with an autoimmune component, such as MS, rheumatoid arthritis, IBS, or IBD
* History of malignancy or any gastrointestinal tract surgery

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All patients were included according to the inclusion and exclusion criteria
Sampling Method: Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2017-12-23 (Actual); Primary Completion 2019-12 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Transcriptional changes in oral microbiota | Baseline, 3 months, 6 months, 9 months, 12 months
  The microbiota measured by 16S rRNA gene

SECONDARY OUTCOMES:
Serum thyroid function changed | Baseline, 3 months, 6 months, 9 months, 12 months
  Serum thyroid function measured by Immunohistochemistry

OTHER OUTCOMES:
Serum thyroid related antibodies changed | Baseline, 3 months, 6 months, 9 months, 12 months
  Serum thyroid related antibodies measured by Immunohistochemistry

CONTACTS AND LOCATIONS:
Overall Officials: Yunwei Wei, Study Director — First Affiliated Hospital of Harbin Medical University
Locations (1):
- First affiliated hospital of Harbin medical university, Harbin, Heilongjiang, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Qin J, Li R, Raes J, Arumugam M, Burgdorf KS, Manichanh C, Nielsen T, Pons N, Levenez F, Yamada T, Mende DR, Li J, Xu J, Li S, Li D, Cao J, Wang B, Liang H, Zheng H, Xie Y, Tap J, Lepage P, Bertalan M, Batto JM, Hansen T, Le Paslier D, Linneberg A, Nielsen HB, Pelletier E, Renault P, Sicheritz-Ponten T, Turner K, Zhu H, Yu C, Li S, Jian M, Zhou Y, Li Y, Zhang X, Li S, Qin N, Yang H, Wang J, Brunak S, Dore J, Guarner F, Kristiansen K, Pedersen O, Parkhill J, Weissenbach J; MetaHIT Consortium; Bork P, Ehrlich SD, Wang J. A human gut microbial gene catalogue established by metagenomic sequencing. Nature. 2010 Mar 4;464(7285):59-65. doi: 10.1038/nature08821. PMID 20203603
- [Background] Dewhirst FE, Chen T, Izard J, Paster BJ, Tanner AC, Yu WH, Lakshmanan A, Wade WG. The human oral microbiome. J Bacteriol. 2010 Oct;192(19):5002-17. doi: 10.1128/JB.00542-10. Epub 2010 Jul 23. PMID 20656903
- [Background] Kabouridis PS, Pachnis V. Emerging roles of gut microbiota and the immune system in the development of the enteric nervous system. J Clin Invest. 2015 Mar 2;125(3):956-64. doi: 10.1172/JCI76308. Epub 2015 Mar 2. PMID 25729852